CLINICAL TRIAL: NCT05901064
Title: Economic Comparison Between the Use of Ultrasonic Scissors and Diathermy for Axillary Clearance in Breast Cancer Patients
Brief Title: Evaluation of Ultrasonic Scissors and Diathermy for Axillary Clearance in Breast Cancer Patients
Acronym: SEROM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, CLuberth, Principal Investigator, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LinkoepingU
Record Dates: First submitted 2023-05-11; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Seroma
Keywords: Seroma; Axillary dissection; Complications
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Intervention Model Description: Double blinded randomized prospective study
Who Masked: Participant, Care Provider
Masking Description: Neither the patients nor the health care providers know with whitch device (Harmonic Focus or diathermy) the patient will be operated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Harmonic Focus (Active Comparator): Patients that are operated with Harmonic Focus
  Interventions: Procedure: Axillary clearance
- Diathermy (Active Comparator): Patients that are operated with conventional diathermy
  Interventions: Procedure: Axillary clearance

INTERVENTIONS:
Procedure: Axillary clearance — Evaluating the use of Harmonic Focus in axillary clearance due to metastasis of breast cancer in axilla
  Other Names: Axillary dissection

SUMMARY:
Breast surgery plays an important role in the treatment of breast cancer. This study investigates if the use of Harmonic Focus has advantages than the use of conventional diathermy in axillary clearance due to metastatic breast cancer.

DETAILED DESCRIPTION:
Breast surgery plays an important role in the treatment of breast cancer. Sometimes cancer cells can spread to lymph nodes in the axill. The first lymph node affected in the armpit is called the sentinel node. Surgery to remove this node can answer the question of whether the cancer has spread to the axill. If the node is affected, further surgery is performed to remove most of the lymph nodes in the armpit, a so-called axillary clereance.

The breast unit at Linköping University Hospital performs about 60 axillary clereance per year. Axillary clereance is associated with a number of complications, such as infections, bleeding, pain, loss of sensation and limited mobility in the arm.

Accumulation of wound fluid in the surgical area is common, affecting about a quarter of patients undergoing surgery. Small amounts of wound fluid usually do not require treatment, but larger accumulations usually require drainage. Patients who have symptoms from armpit wound fluid have to make repeated return visits so that a nurse drains the fluid using a needle. This poses several risks to the patient such as infection and/or bleeding. This, in turn, can delay the start of additional treatment and can put a financial burden on both the patient and the healthcare system.

Today, the investigators use a device with a weak electric current (diathermy) to remove lymph nodes from the armpit. Harmonic Focus ® is a pair of scissors that instead uses ultrasound waves to divide the tissue. There are scientific studies showing that the use of ultrasonic scissors reduces the risk of fluid accumulation and thus the risk of complications after surgery[1, 2]. The investigators want to conduct a prospective study, an economic analysis comparing the costs of using diathermy versus Harmonic Focus®.

In addition, patients will complete a quality of life questionnaire before surgery, approximately 4-6 weeks after and one year after surgery. The results of the questionnaires will be compared between the Harmonic Focus® and the diathermy group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* All patients who will undergo axillary evacuation
* Informed consent

Exclusion Criteria:

* Patients who have previously undergone axillary evacuation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Economic comparison between the use of ultrasonic scissors and diathermy for axillary dissection in breast cancer patients. | 12 months
  Unit of measures: Costs of extra visits with nurse, physiotherapist or surgeon, antibiotics, PICO, re-interventions due to complications, microbiological cultures, incapacity to work, hospitalizations

SECONDARY OUTCOMES:
Function before and after breast cancer treatment. Lymph-ICF Survey | 12 months
  Questionnaire
Complication frequency between the use of ultrasonic scissors and diathermy for axillary | 12 months
  Comlplication frequency comparison

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Linkoping, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bohm D, Kubitza A, Lebrecht A, Schmidt M, Gerhold-Ay A, Battista M, Stewen K, Solbach C, Kolbl H. Prospective randomized comparison of conventional instruments and the Harmonic Focus((R)) device in breast-conserving therapy for primary breast cancer. Eur J Surg Oncol. 2012 Feb;38(2):118-24. doi: 10.1016/j.ejso.2011.11.003. Epub 2011 Dec 5. PMID 22152942
- [Background] Faisal M, Fathy H, Shaban H, Abuelela ST, Marie A, Khaled I. A novel technique of harmonic tissue dissection reduces seroma formation after modified radical mastectomy compared to conventional electrocautery: a single-blind randomized controlled trial. Patient Saf Surg. 2018 May 17;12:8. doi: 10.1186/s13037-018-0155-3. eCollection 2018. PMID 29796089
- [Background] Giuliano AE, Hunt KK, Ballman KV, Beitsch PD, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, McCall LM, Morrow M. Axillary dissection vs no axillary dissection in women with invasive breast cancer and sentinel node metastasis: a randomized clinical trial. JAMA. 2011 Feb 9;305(6):569-75. doi: 10.1001/jama.2011.90. PMID 21304082
- [Background] Galimberti V, Cole BF, Zurrida S, Viale G, Luini A, Veronesi P, Baratella P, Chifu C, Sargenti M, Intra M, Gentilini O, Mastropasqua MG, Mazzarol G, Massarut S, Garbay JR, Zgajnar J, Galatius H, Recalcati A, Littlejohn D, Bamert M, Colleoni M, Price KN, Regan MM, Goldhirsch A, Coates AS, Gelber RD, Veronesi U; International Breast Cancer Study Group Trial 23-01 investigators. Axillary dissection versus no axillary dissection in patients with sentinel-node micrometastases (IBCSG 23-01): a phase 3 randomised controlled trial. Lancet Oncol. 2013 Apr;14(4):297-305. doi: 10.1016/S1470-2045(13)70035-4. Epub 2013 Mar 11. PMID 23491275
- [Background] de Boniface J, Frisell J, Andersson Y, Bergkvist L, Ahlgren J, Ryden L, Olofsson Bagge R, Sund M, Johansson H, Lundstedt D; SENOMAC Trialists' Group. Survival and axillary recurrence following sentinel node-positive breast cancer without completion axillary lymph node dissection: the randomized controlled SENOMAC trial. BMC Cancer. 2017 May 26;17(1):379. doi: 10.1186/s12885-017-3361-y. PMID 28549453
- [Background] Sowa Y, Numajiri T, Kawarazaki A, Sakaguchi K, Taguchi T, Nishino K. Preventive effects on seroma formation with use of the harmonic focus shears after breast reconstruction with the latissimus dorsi flap. J Plast Surg Hand Surg. 2016 Dec;50(6):349-353. doi: 10.1080/2000656X.2016.1178129. Epub 2016 May 5. PMID 27146859
- [Background] Selvendran S, Cheluvappa R, Tr Ng VK, Yarrow S, Pang TC, Segara D, Soon P. Efficacy of harmonic focus scalpel in seroma prevention after axillary clearance. Int J Surg. 2016 Jun;30:116-20. doi: 10.1016/j.ijsu.2016.04.041. Epub 2016 Apr 29. PMID 27142863
- [Background] Hung SH, Chu D, Chen FM, Chen T, Chen RC. Evaluation of the harmonic scalpel in breast conserving and axillary staging surgery. J Chin Med Assoc. 2012 Oct;75(10):519-23. doi: 10.1016/j.jcma.2012.07.006. Epub 2012 Sep 15. PMID 23089404
- [Background] He Q, Zhuang D, Zheng L, Fan Z, Zhou P, Zhu J, Lv Z, Chai J, Cao L. Harmonic focus versus electrocautery in axillary lymph node dissection for breast cancer: a randomized clinical study. Clin Breast Cancer. 2012 Dec;12(6):454-8. doi: 10.1016/j.clbc.2012.07.014. Epub 2012 Oct 3. PMID 23040644